CLINICAL TRIAL: NCT06112782
Title: Efficacy and Safety of Keravive by Hydrafacial for Scalp Health and Enhanced Hair Quality in Patients With Androgenic Alopecia a Take-Home Hair Care Product and an In-Clinic Scalp Stimulating Treatment
Brief Title: Keravive by Hydrafacial for Scalp Health and Enhanced Hair Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beauty Health (Industry)
Collaborators: Skin Surgery Medical Group (Other); ATS Clinical Research (Other); Callender Center for Clinical Research (Other); Rebecca Fitzgerald MD Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HF-1801
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Keravive by Hydrafacial Treatment (Other): Subjects will receive 3 in-office scalp Keravive by Hydrafacial treatments every 4 weeks in combination with daily application of Keravive Peptide Spray.
  Interventions: Device: Keravive by Hydrafacial Treatments

INTERVENTIONS:
Device: Keravive by Hydrafacial Treatments — Scalp hydradermabrasion

SUMMARY:
The study aims to assess the efficacy and safety of Keravive by Hydrafacial treatments and Keravive Peptide Spray for scalp health and enhancing hair quality in patients with androgenic alopecia. This study is intended to be a single arm study. Suitable subjects who meet all inclusion criteria and consented will undergo 3 in-office Keravive by Hydrafacial treatments at Day 0 and Weeks 4 and 8 in combination with daily application on Keravive Peptide Spray at home.

Subjects will be assessed at Day 0, and Weeks 4, 8, and 20 by investigators using the Norwood Scale (males), Ludwig Classification (females), and a series of Likert scales for ranking improvement in scalp health and hair quality.

DETAILED DESCRIPTION:
This study is intended to be a single arm study. Suitable subjects who meet all inclusion criteria and consented will undergo 3 in-office Keravive by Hydrafacial treatments at baseline and Weeks 4 and 8 in combination with daily application on Keravive Peptide Spray at home.

Subjects will be assessed at baseline, and Weeks 4, 8, and 20 by investigators using the Norwood Scale (males), Ludwig Classification (females), and a series of Likert scales for ranking improvement in scalp health and hair quality.

Efficacy will be assessed through a series of dynamic and static questionnaires. Investigators will complete static questionnaires at Day 0 and Weeks 4, 8 and 20 rating the subjects' hair appearance, thinning, and temporal line recession using Likert scales. Subjects will complete dynamic questionnaires at Weeks 4, 8 and 20 to compare their current state to their baseline condition for scalp symptoms (itchiness, dryness, and flakiness) and hair quality (overall health, fullness, evenness, pigment, hair growth, and hair loss) using Likert scales. Subjects will also rank their hair appearance at Day 0, Week 4, 8, and 20. Photography will be performed at each study visit. Safety assessments will include investigator- and subject-reported adverse events (AEs) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Norwood Scale score of 2, 3 or 3 Vertex (males) and Ludwig Classification of Type I-1, I-2 or I-3 (females).

Exclusion Criteria:

* Non-study hair loss treatments (e.g., dutasteride, finasteride, minoxidil, nutraceuticals, PRP therapy, laser or LED scalp treatments, etc.)
* Salon treatments such as straightening, perms or coloring.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Hair Thinning and Temporal Hairline Recession | Day 0, Weeks 4, 8, and 20
  Investigator assessments of hair thinning and temporal line recession using Likert scales.
Scalp Health | Weeks 4, 8, and 20
  Subject-assessed improvement in scalp itchiness, dryness, and flakiness using Likert scales.
Hair Appearance | Day 0, Weeks 4, 8, and 20
  Investigator and subject assessments of hair appearance using Likert scales.

SECONDARY OUTCOMES:
Hair Health | Weeks 4, 8, and 20
  Subject-assessed improvement in hair health, fullness, evenness, pigment, hair growth and loss using Likert scales.

OTHER OUTCOMES:
Adverse Events | 20 weeks
  Incidence and severity of investigator and subject reports of adverse events.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rebecca Fitzgerald MD Inc, Los Angeles, California
  - Laser & Skin Surgery Medical Group, Inc, Sacramento, California
  - ATS Clinical Research, Santa Monica, California
  - Callender Center for Clinical Research, Glenn Dale, Maryland

IPD SHARING:
Plan to Share IPD: No
Plan for data to be published in peer-reviewed journal and presented at conferences.